CLINICAL TRIAL: NCT02870192
Title: Intra-operative Adverse Events During Laparoscopic Ventral Mesh Rectopexy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Pierpaolo Sileri, Prof, University of Rome Tor Vergata
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 91/12
Record Dates: First submitted 2016-08-09; First posted 2016-08-17 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Rectal Prolapse
Keywords: Rectal Prolapse
MeSH Terms: conditions — Rectal Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rectal Prolapse (Experimental): Patients with rectal prolapse, who will underwent laparoscopic ventral mesh rectopexy. The implemented mesh may be synthetic or biological.
  Interventions: Procedure: Laparoscopic ventral mesh rectopexy

INTERVENTIONS:
Procedure: Laparoscopic ventral mesh rectopexy — Laparoscopic opening of the Daglous pouch, dissection till reach the levator ani muscle, mesh implementation and fixation, closure of the daglous. The mesh implemented may be synthetic or biological mesh.

SUMMARY:
Outcomes of laparoscopic ventral mesh rectopexy are well known, but data on intra-operative adverse events is scant. A multicenter pool-analysis of prospectively collected database on 1384 patients with internal/external rectal prolapse toke place. Overall 72 (5%) patients experienced complications, 41 discovered and managed intraoperatively, 22 postoperative complications, and 9 required readmission. Despite accepted lower rate of morbidity, these results come from four well equipped European centers by four surgeons practiced at least 200 LVMR.

DETAILED DESCRIPTION:
Multicenter pooled-analysis of LVMR for internal/external rectal prolapse. All events occurred and discovered intra-operatively or passed undiagnosed and appeared within 30-days postoperatively (same admission/readmission) will included, with classification according to the Clavien-Dindo classification.

ELIGIBILITY:
Inclusion Criteria:

* all patients underwent laparoscopic ventral mesh rectopexy for internal and external rectal prolapse

Exclusion Criteria:

* other condition than rectal prolapse

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-06 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
intra-operative complications | 30 days postoperative
  All complications occur during the operation and discovered and managed during the operation or passed undiscovered and discovered postoperative during the same admission or require readmission

CONTACTS AND LOCATIONS:
Overall Officials: Pierpaolo Sileri, MD, PhD, Principal Investigator — University of Rome Tor Vergata

IPD SHARING:
Plan to Share IPD: Undecided